CLINICAL TRIAL: NCT03765944
Title: A Single Dose, Randomized, Open-label, 2-Period, 2-way Crossover, Bioequivalence Study of Sirolimus Granules and Sirolimus Tablets in Japanese Healthy Adults
Brief Title: Bioequivalence Study of NPC-12 (Sirolimus) Granules and Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NPC-12T-1
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Bioequivalence Study
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPC-12 granule (Active Comparator): NPC-12 granules (1.0g: 2mg sirolimus)
  Interventions: Drug: sirolimus
- NPC-12T tablet (Active Comparator): NPC-12T 2 tablets (2mg sirolimus)
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — SIngle administration under fasted condition

SUMMARY:
The purpose of this study is to evaluate the bioequivalece of NPC-12 granules in compare with NPC-12T tablets in Japanese healthy Adults

ELIGIBILITY:
Inclusion Criteria:

1. Japanese healthy subjects aged 20 to 39 years of age
2. Subjects with BMI ≥ 18.5 kg/m2 and < 25.0 kg/m2
3. Subjects who are considered by the investigator as suitable for participation in the trial from lab test results at screening
4. Subjects who are considered by the investigator as suitable for participation in the trial from lab test results on the day before administration
5. Subjects who write informed consent
6. Subjects who are able to comply with the study requirements during the study period

Exclusion Criteria:

1. Subjects who have a history of hypersensitivity to sirolimus or sirolimus derivative
2. Subjects who have a history of hypersensitivity or allergies to other drug
3. SUbjects who have an acute or chronic infectious diseases
4. Subjects who have a current or a history of disease which is considered inappropriate to be involved in the study, or who has any current disease to require treatments
5. Subjects who have diagnosed with alcoholism or a history of alcoholism
6. Subjects who have an abnormal findings (pneumonia, etc) from the result of chest CT at screening
7. Subjects who have been administered other investigational drug within 12 weeks before the initial administration
8. Subjects who have performed blood collection or donation as follows

   * Collected or donated 200 ml or more whole blood within 4 weeks before the initial administration
   * Male subject; collected or donated more than 400 mL whole blood within 12 weeks before the initial administration
   * Female subjects; collected or donated more than 400 mL whole blood within 16 weeks before the initial administration
   * Collected or donated blood component within 2 weeks before the initial administration
9. Subjects who have positive results for HBs antigen, HBs antibody, HBc antibody, HCV antibody, HIV antigen/antibody, or syphilis
10. Subjects who received any non-prescription or prescription drug within 12 weeks before the initial administration
11. Subjects who are pregnant/lactating, or do not agree to contraception during the period from the screening until 8 weeks after the final administration due to planning to become pregnant
12. Subjects who cannot speak, read and write in Japanese
13. Subjects who are considered by the investigator as unsuitable for participation in the trial

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2018-12-29 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
Blood sirolimus concentration | Pre-dose and post-dose (0.5, 1, 1.5, 2, 4, 8, 12, 18, 24, 48 and 72 hours)
  Whole blood concentration of sirolimus will be measured and compared between NPC-12 granules and NPC-12T tablets.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Soigner, Matsudo, Chiba, Japan

IPD SHARING:
Plan to Share IPD: No